CLINICAL TRIAL: NCT05461131
Title: A Phase 2b, Placebo-Controlled, Randomized Study of BPZE1 Intranasal Pertussis Vaccine in Healthy Adults to Assess Protection Against Colonization Following Challenge With Virulent Wild-Type Bordetella Pertussis
Brief Title: Pertussis Challenge Study in Adults Vaccinated With BPZE1
Acronym: CHAMPION-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ILiAD Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IB-202P
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Results first posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Pertussis/Whooping Cough; Bordetella Pertussis, Whooping Cough
Keywords: Bordetella Pertussis; BPZE1; Vaccine; Live Attenuated Vaccine; Challenge Study
MeSH Terms: conditions — Whooping Cough | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BPZE1 (Experimental): Participants will receive an intranasal dose of BPZE1 via the mucosal atomization device followed by a dose of the challenge strain (B. Pertussis strain 1917) approximately 60-120 days later. Participants will receive azithromycin for 3 days beginning 14 days after administration of the challenge strain.
  Interventions: Biological: BPZE1; Drug: Azithromycin; Other: Bordetella Pertussis Challenge Strain
- Placebo (Placebo Comparator): Participants will receive an intranasal dose of placebo via the mucosal atomization device followed by a dose of the challenge strain (B. Pertussis strain 1917) approximately 60-120 days later. Participants will receive azithromycin for 3 days beginning 14 days after administration of the challenge strain.
  Interventions: Biological: Placebo; Drug: Azithromycin; Other: Bordetella Pertussis Challenge Strain

INTERVENTIONS:
Biological: BPZE1 — Live attenuated vaccine
  Arms: BPZE1
Biological: Placebo — Placebo
  Arms: Placebo
Drug: Azithromycin — Antibiotic
Other: Bordetella Pertussis Challenge Strain — Challenge Strain

SUMMARY:
This is a randomised, double-blinded, placebo-controlled trial of BPZE1 that includes virulent B. pertussis challenge followed by a safety follow-up.

DETAILED DESCRIPTION:
This Phase 2b challenge study will investigate colonisation rates, immunologic response, and the safety of BPZE1 vaccination to potentially protect against colonising, virulent wild-type B. pertussis infection in healthy adults using a virulent challenge model. Consenting, eligible participants will receive a single dose of BPZE1 or placebo. 2-4 months later they will be challenged with B. pertussis and admitted to a challenge unit. Participants will remain in the challenge unit for a total of 17 days and 16 nights during which time they will be monitored closely. If a participant develops symptoms of pertussis (per investigator discretion), antibiotic (azithromycin) will be started and the participant will remain in the unit for 3 additional days of observation before discharge. If symptoms of pertussis do not develop, then participants will receive antibiotic (azithromycin) from Days 14-16 of the challenge unit stay. Participants will undergo safety follow-up for at least 6 months post-vaccination and at least 3 months post-challenge, for a total follow-up of 6-7 months.

ELIGIBILITY:
Key Inclusion Criteria:

1. Correctly answer all questions in the questionnaire provided during the consent process to ensure understanding of the study
2. Willing to refrain from any nasal sprays (including intranasal steroid sprays) and nasal washes not part of the study for 14 days prior to vaccination (Day 0) and for 28 days following vaccination and challenge
3. Non-smoker at the time of enrolment, has not smoked (or vaped) in the past 7 days prior to vaccination (including marijuana), and is willing not to smoke (or vape; including marijuana) from the time of vaccination throughout the challenge unit phase
4. Sufficiently vaccinated (per site and local guidelines) against severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2; proof of vaccination required) >14 days prior to study vaccination
5. Able to understand and comply with planned study procedures including admission for virulent challenge for 17 days and willingness to take the curative antibiotic regimen (azithromycin after inoculation with B. pertussis)
6. Willing to provide written agreement to and abide by infection control rules from challenge until 1 week following completion of azithromycin eradication

Exclusion Criteria:

1. Body mass index <17 or >30 kg/m2
2. History of being vaccinated against pertussis within 5 years of enrolment
3. History of never being vaccinated for pertussis in lifetime
4. A diagnosis of pertussis by laboratory confirmation or by physician diagnosis in the past 5 years
5. Previously participated in a pertussis challenge study
6. Screening laboratory values outside of the normal ranges
7. Existing chronic disorders of lung, kidney, heart, liver, diabetes, immunodeficiency, autoimmune or significant neurologic condition
8. Use of illicit drugs (excluding marijuana), evidenced by urine toxicology at Screening or a history of drug/alcohol abuse within the past 2 years
9. History of active cancer (malignancy) in the last 10 years (except for adequately treated non-melanomatous skin carcinoma)
10. History of Guillain-Barré syndrome (genetic/congenital or acquired)
11. History of head trauma with potential of cribriform plate fracture within 1 year prior to Day 0
12. History of nasal or sinus surgery within 6 months or receipt of facial cosmetic fillers within 3 months prior to Day 0 or diagnosis of nasal polyps
13. Received immunosuppressive therapy or other immune-modifying drugs (including but not limited to systemic corticosteroids, biologics and methotrexate) in the past 6 months, is on scheduled immunosuppressive therapy or is planning to start immunosuppressive therapy during the trial.
14. Received immunoglobulins or any blood products within 3 months prior to study vaccine administration or planned receipt during the study
15. Lives in the same home or has routine contact (face to face <2 meters) with persons with known immunodeficiency including persons on immunosuppressant therapy, from study vaccination to challenge and for 1 week after exiting the challenge unit
16. Resides in the same home, works regularly with, or has contact (face to face <2 meters), with infants less than 1 year of age, partially immunised infants or pregnant women, adults >65 years of age who have not received a dose of acellular pertussis vaccine (e.g. Tdap) within the past 10 years from study vaccination to challenge and for 1 week after exiting the challenge unit
17. Known hypersensitivity to any component of the study vaccine
18. Contraindications or allergic to azithromycin, erythromycin or other macrolide antibiotics
19. Taking medication that may interact with azithromycin (e.g., nelfinavir, warfarin, digoxin and phenytoin)
20. Inability to adhere to the protocol, visit schedule or sample collection needs (including housing in the challenge unit)
21. Participation in any other clinical trial for the testing of an unlicensed product during the previous 3 months or planned during the study conduct

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Oxford Vaccine Group, Oxford
  - University Hospital Southampton, Southampton

REFERENCES:
- [Derived] Gbesemete D, Ramasamy MN, Ibrahim M, Hill AR, Raud L, Ferreira DM, Guy J, Dale AP, Laver JR, Coutinho T, Faust SN, Reed TAN, Babbage G, Weissfeld L, Lang W, Locht C, Samal V, Goldstein P, Solovay K, Rubin K, Noviello S, Read RC. Efficacy, immunogenicity, and safety of the live attenuated nasal pertussis vaccine, BPZE1, in the UK: a randomised, placebo-controlled, phase 2b trial using a controlled human infection model with virulent Bordetella pertussis. Lancet Microbe. 2025 Dec;6(12):101211. doi: 10.1016/j.lanmic.2025.101211. Epub 2025 Dec 1. PMID 41344352

RESULTS

PARTICIPANT FLOW:
Groups:
- BPZE1: Participants will receive an intranasal dose of BPZE1 via the mucosal atomization device followed by a dose of the challenge strain (B. pertussis strain 1917) approximately 60-120 days later. Participants will receive azithromycin for 3 days beginning 14 days after administration of the challenge strain.
  BPZE1: Live attenuated B. pertussis vaccine
  Azithromycin: Antibiotic
  Bordetella Pertussis strain 1917 Challenge: Challenge Strain
- Placebo: Participants will receive an intranasal dose of placebo via the mucosal atomization device followed by a dose of the challenge strain (B. pertussis strain 1917) approximately 60-120 days later. Participants will receive azithromycin for 3 days beginning 14 days after administration of the challenge strain.
  Placebo: Placebo
  Azithromycin: Antibiotic
  Bordetella Pertussis strain 1917 Challenge: Challenge Strain
Period: Overall Study
Arm/Group | BPZE1 | Placebo
Started | 26 | 27
Challenged With Virulent B. Pertussis | 24 (Reasons for Subjects Not Challenged (n=2): * 1 subject moved out of country * 1 subject unable to challenge for personal reasons) | 22 (Reasons for Subjects Not Challenged (n=5): * 2 subjects discontinued from the study before challenge * 2 subjects were lost to follow-up * 1 subject experienced an unrelated AE)
Completed | 26 | 25
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BPZE1 | Placebo | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 27 | 53
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.3 (7.77) | 31.4 (9.16) | 30.4 (8.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 12 | 14 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Colonized Following Virulent Challenge
Description: Participants by treatment group (BPZE1 and placebo) colonized on any day (Challenge Day 9, 11 or 14) following virulent challenge as determined by culture.
Time Frame: Challenge Day 9, 11 or 14
Population: Subjects who received an adequate inoculum defined prospectively as challenge dose >=0.5x10^5 CFU were evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 20 | 16
Participants | 8 | 12

2. Secondary Outcome: GMFR of Mucosal Anti-pertussis S-IgA Antibody
Description: The geometric mean fold rise (GMFR) of mucosal anti-pertussis S-IgA antibody (whole cell extract [WCE], FHA, PRN, PT and fimbriae types 2 and 3 [FIM2/3]) from baseline to Day 28 (BPZE1 and placebo). Secretory IgA to be normalized ([specific S-IgA]/[total S-IgA])
Time Frame: Day 28
Population: Available baseline and Day 28 samples
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Rise
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 25
Geometric Mean Fold Rise
  WCE | 3.2 [2.1 to 4.7] | 1.0 [0.8 to 1.3]
  FHA | 5.0 [3.0 to 8.2] | 1.1 [0.8 to 1.5]
  PRN | 5.3 [2.9 to 9.8] | 1.0 [0.7 to 1.3]
  PT | 1.7 [1.2 to 2.5] | 1.2 [0.9 to 1.6]
  FIM 2/3 | 9.1 [4.9 to 16.9] | 1.1 [0.9 to 1.4]

3. Secondary Outcome: GMFR of Serum IgA Antibody
Description: The GMFR of serum IgA antibody (WCE, FHA, PRN, PT and FIM2/3) from baseline to Day 28 (BPZE1 and placebo)
Time Frame: Day 28
Population: Available baseline and Day 28 samples
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Rise
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 25
Geometric Mean Fold Rise
  WCE | 2.6 [1.9 to 3.4] | 1.2 [1.0 to 1.4]
  FHA | 3.0 [2.2 to 4.0] | 1.1 [1.0 to 1.3]
  PRN | 3.7 [2.2 to 6.2] | 1.0 [0.9 to 1.1]
  PT | 1.5 [1.1 to 2.0] | 1.1 [1.0 to 1.3]
  FIM 2/3 | 5.0 [3.1 to 8.2] | 1.0 [1.0 to 1.1]

4. Secondary Outcome: GMFR of Serum IgG Antibody
Description: The GMFR of serum IgG antibody (WCE, FHA, PRN, PT and FIM2/3) from baseline to Day 28 (BPZE1 and placebo)
Time Frame: Day 28
Population: Available baseline and Day 28 samples
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Fold Rise
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 25
Geometric Mean Fold Rise
  WCE | 1.5 [1.3 to 1.7] | 1.1 [1.0 to 1.1]
  FHA | 1.7 [1.2 to 2.2] | 1.0 [0.8 to 1.2]
  PRN | 3.1 [1.9 to 5.0] | 1.1 [0.8 to 1.5]
  PT | 2.1 [1.4 to 3.0] | 1.0 [0.7 to 1.3]
  FIM 2/3 | 2.9 [1.9 to 4.5] | 0.9 [0.7 to 1.2]

5. Secondary Outcome: Safety: Number of Participants With Solicited AEs for Reactogenicity
Description: Occurrence and intensity of solicited AEs for nasal/respiratory and systemic reactogenicity through 7 days following vaccination by treatment group (BPZE1 and placebo)
Time Frame: Day 7
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 27
Participants
  Nasal/Respiratory | 17 | 20
  Systemic | 18 | 16

6. Secondary Outcome: Safety: Number of Participants With Treatment Emergent Adverse Events
Description: Occurrence and intensity of TEAEs through 28 days following study vaccination and following challenge by treatment group (BPZE1 and placebo)
Time Frame: Day 28
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 27
Participants | 7 | 9

7. Secondary Outcome: Safety: Number of Participants With TEAEs Related to Vaccination or Related to Challenge
Description: Occurrence and intensity of TEAEs related to vaccination from time of vaccination to challenge or related to challenge for 3 months after challenge by treatment group (BPZE1 and placebo)
Time Frame: Day 60-120 post vaccination and Day 90 post challenge
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 27
Participants | 4 | 8

8. Secondary Outcome: Safety: Number of Participants With AESI and SAE
Description: Occurrence, intensity, and relationship to study vaccine of AESIs and SAEs from vaccination through end of study (EOS) by treatment group (BPZE1 and placebo)
Time Frame: Day 180
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | BPZE1 | Placebo
Number analyzed (Participants) | 26 | 27
Participants
  AESI (COVID-19) | 0 | 1
  SAE | 0 | 0

ADVERSE EVENTS:
Time Frame: SAEs and deaths collected through end of study - up to 7 months. Unsolicited AEs collected up to 28 days post-vaccination and 28 days post-challenge.
Arm/Group | BPZE1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 7/26 | 9/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BPZE1 (N=26) | Placebo (N=27)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Other (General disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT05461131/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT05461131/SAP_001.pdf